CLINICAL TRIAL: NCT03365102
Title: Modulating Impulsivity in Suicidal Adolescents With tDCS: A Proof of Concept Study
Brief Title: Modulating Impulsivity in Suicidal Adolescents With Transcranial Direct Current Stimulation (tDCS)
Acronym: tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Richard Liu, Assistant Professor, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Liu 002017
Record Dates: First submitted 2017-08-02; First posted 2017-12-07 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Impulsive Behavior
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Intervention Model Description: anodal tDCS over the rIFG, anodal tDCS over the lOFC, sham stimulation condition
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither participant or outcome aware of condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- anodal tDCS over the rIFG, (Experimental): anodal tDCS over the rIFG,
  Interventions: Device: anodal tDCS over the rIFG,
- anodal tDCS over the lOFC (Experimental): anodal tDCS over the lOFC
  Interventions: Device: anodal tDCS over the lOFC,
- sham tDCS stimulation (Placebo Comparator): sham tDCS stimulation
  Interventions: Device: sham tDCS stimulation condition

INTERVENTIONS:
Device: anodal tDCS over the rIFG, — tDCS at a constant current of 1.5 milliampere (mA) will be applied for one 20-minute session over the right inferior frontal gyrus . Resting-state EEG for 10 minutes will be recorded immediately prior to and after tDCS. After post-tDCS resting state EEG is acquired, EEG is recorded to extract Evoked Response Potentials in a single-blind procedure. The participants and assessors will be blind to experimental condition.
  Arms: anodal tDCS over the rIFG,
Device: anodal tDCS over the lOFC, — tDCS at a constant current of 1.5 mA will be applied for one 20-minute session over the left orbitofrontal cortex . Resting-state EEG for 10 minutes will be recorded immediately prior to and after tDCS. After post-tDCS resting state EEG is acquired, EEG is recorded to extract Evoked Response Potentials in a single-blind procedure. The participants and assessors will be blind to experimental condition.
  Arms: anodal tDCS over the lOFC
Device: sham tDCS stimulation condition — In the sham condition, the current will be ramped up to 1.5 mA for 30 seconds and then ramped back down to 0. As this commonly used sham procedure produces a brief tingling sensation, participants are kept unaware of their experimental condition. Resting-state EEG for 10 minutes will be recorded immediately prior to and after the sham tDCS. After post-sham stimulation resting state EEG is acquired, EEG is recorded to extract Evoked Response Potentials in a single-blind procedure. The participants and assessors will be blind to experimental condition.
  Arms: sham tDCS stimulation

SUMMARY:
As a first step toward investigating whether modulation of impulsivity and associated neural pathways may yield clinically meaningful changes in risk for adolescent suicidal behavior, the R21 is a proof-of concept study evaluating the potential for tDCS targeting brain regions associated with behavioral impulsivity (right inferior frontal gyrus [rIFG]) and cognitive impulsivity (left orbitofrontal cortex [lOFC]) to modulate these facets of impulsivity in a sample of adolescent suicide attempters. Participants will be randomly assigned to receive anodal tDCS over the rIFG, anodal tDCS over the lOFC, or a sham stimulation condition, in a three-group design. Task-based measures of behavioral and cognitive impulsivity will be administered before and after tDCS or sham stimulation. Additionally, electroencephalography (EEG) and event-related potential (ERP) data will be collected during the impulsivity tasks, and resting-state EEG data will be collected pre- and post-tDCS administration to confirm engagement of the targeted brain regions and to delineating the neural pathways underlying the effects of tDCS on impulsivity.

DETAILED DESCRIPTION:
Suicide is one of the leading causes of death in adolescence. To improve the ability to predict and prevent suicidal behavior, there is a pressing need for research in this area to advance beyond identifying risk factors toward a greater focus on the mechanisms of risk for this behavior. In particular, elucidating the neural pathways underlying risk for suicidal behavior is important insofar as such work may yield specific and modifiable targets for clinical intervention. The adoption of new experimental paradigms providing experimental control over potentially modifiable risk factors has been recommended as a means of meaningfully advancing the field in this regard. Although yet to be applied to the study of suicidality, transcranial direct current stimulation (tDCS), in conjunction with measures of electroencephalography (EEG) and event-related potentials (ERPs), may hold promise as an experimental paradigm in the study of potentially modifiable risk factors, and underlying neural mechanisms, for suicidality. One such risk factor of particular relevance to suicide in adolescence is state-sensitive aspects of impulsivity. Impulsivity has been consistently linked with suicidality, with this association appearing to be stronger in adolescence than adulthood. As a first step toward investigating whether modulation of impulsivity and associated neural pathways may yield clinically meaningful changes in risk for adolescent suicidal behavior, the R21 is a proof-of concept study evaluating the potential for tDCS targeting brain regions associated with behavioral impulsivity (right inferior frontal gyrus [rIFG]) and cognitive impulsivity (left orbitofrontal cortex [lOFC]) to modulate these facets of impulsivity in a sample of adolescent suicide attempters. Participants will be randomly assigned to receive anodal tDCS over the rIFG, anodal tDCS over the lOFC, or a sham stimulation condition, in a three-group design. Task-based measures of behavioral and cognitive impulsivity will be administered before and after tDCS or sham stimulation. Additionally, EEG and ERP data will be collected during the impulsivity tasks, and resting-state EEG data will be collected pre- and post-tDCS administration to confirm engagement of the targeted brain regions and to delineating the neural pathways underlying the effects of tDCS on impulsivity.

ELIGIBILITY:
Inclusion Criteria:

* have attempted suicide prior to admission
* speak and read English fluently
* do not display evidence of significant cognitive impairment, based on a standard psychiatric exam as well as school records on admission
* are not actively psychotic at time of intake.

Exclusion Criteria:

* a significant general medical condition
* history of seizure, head injury, brain surgery or tumor
* intracranial metallic implants or implanted electrical devices
* substance abuse or dependence in the past six months.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Liu, PhD, Principal Investigator — Lifespan
Locations (1):
- Bradley Hospital, Riverside, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Analysis files will be constructed from the stored electronic data and will be stripped of identifying information with the Safe Harbor method. Specifically, youth and their parents will be identified with a family identifier and person identifier number that is randomly generated and not related to any element of their personal identifying information. No names, addresses, telephone numbers, fax numbers, email addresses, social security numbers, medical records, etc. will be retained. Dates will contain only year and a randomly generated day-of-the-year. The investigators will only share it with external investigators when a data use agreement (DUA) is executed between Lifespan and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project, and schedule for data destruction. The data will be made available on April 1, 2021 by the PI
Supporting Information: Study Protocol, ICF
Time Frame: April 1, 2021
Access Criteria: The investigators will only share it with external investigators when a data use agreement (DUA) is executed between the Brown University and the requester's institution. The DUA will specify the requested data elements (each of which must be justified), the specific research question, the timeline for the project, and schedule for data destruction.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anodal tDCS Over the rIFG, | Anodal tDCS Over the lOFC | Sham tDCS Stimulation
Started | 22 | 22 | 20
Completed | 18 | 21 | 19
Not Completed | 4 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data for participants who completed the study procedures are reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal tDCS Over the rIFG, | Anodal tDCS Over the lOFC | Sham tDCS Stimulation | Total
Number analyzed (Participants) | 18 | 21 | 19 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 21 | 19 | 58
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 14 | 45
  Male | 4 | 4 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 2 | 12
  Not Hispanic or Latino | 13 | 16 | 17 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 8
  White | 7 | 12 | 12 | 31
  More than one race | 7 | 6 | 3 | 16
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 21 | 19 | 58
PROMIS Depression [Mean (Standard Deviation); unit: units on a scale] — This is a self-report measure of depressive symptoms. Total scores are reported with higher scores reflecting greater depression. Range of total scores = 8 to 40. Population: 2 participants were missing data.
  units on a scale
    number analyzed (Participants) | 18 | 19 | 19 | 56
    (all) | 49 (10) | 47 (12) | 47 (12) | 47.64285714 (11.22728587)
Conners-3 Self-Report [Mean (Standard Deviation); unit: units on a scale] — The inattention subscale total score ranges from 0-33, with higher scores reflecting greater inattention. The hyperactivity/impulsivity subscale total score ranges from 0-42, with higher scores indicating greater hyperactivity/impulsivity. Population: 3 participants were missing data
  units on a scale
    Inattention subscale: number analyzed (Participants) | 17 | 21 | 18 | 56
    Inattention subscale | 16 (8) | 16 (9) | 15 (8) | 15.67857143 (8.250855918)
    Hyperactivity/impulsivity subscale: number analyzed (Participants) | 17 | 20 | 19 | 56
    Hyperactivity/impulsivity subscale | 14 (7) | 17 (7) | 12 (7) | 14.39285714 (7.191354839)
Stop Signal Task [Mean (Standard Deviation); unit: milliseconds] — The stop signal task produces stop signal response time (SSRT) as the outcome variable in milliseconds, with hypothetically possible scores range from 0 to no hypothetical upper limit. Greater scores reflect greater impulsivity. Population: 6 participants were missing data
  milliseconds
    number analyzed (Participants) | 16 | 18 | 18 | 52
    (all) | 353 (414) | 276 (328) | 233 (247) | 284.8076923 (330.2148165)
Delay discounting task [Mean (Standard Deviation); unit: score on a scale] — This task assessed discounting larger future rewards for smaller immediate ones. The point where a person is equally likely to prefer immediate vs delayed reward (the indifference point) is determined for several and combinations of reward sizes and lengths of time. Area under the curve (AUC) is calculated by summing the results of the following for each delay and indifference point pair: x2-x1[(y1 + y2)/2]. x1 and x2 are successive delays and y1 and y2 are indifference points for those delays. AUC range=0-1. Larger AUCs reflect less impulsivity. Population: 3 participants were missing data
  score on a scale
    number analyzed (Participants) | 17 | 20 | 18 | 55
    (all) | .45 (.3) | .31 (.22) | .5 (.31) | 0.415454545 (0.284301081)

OUTCOME MEASURES:

1. Primary Outcome: Stop Signal Task (SST)
Description: The Stop-Signal Task (SST) is a task requiring inhibition of a prepotent motor response. The SST requires participants to respond to a target stimulus as quickly and accurately as possible by pressing a button, but also to withhold their response when they hear an auditory signal. Thus, this task involves a competition between activating and inhibiting processes. The primary outcome variable is change in the stop signal reaction time (SSRT) for the task administered seconds to minutes before and seconds to minutes after stimulation. The theoretical minimum is zero seconds and there is no theoretical maximum. Higher SSRT scores reflect greater impulsivity.
Time Frame: Within an hour post-stimulation condition
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Anodal tDCS Over the rIFG, | Anodal tDCS Over the lOFC | Sham tDCS Stimulation
Number analyzed (Participants) | 15 | 15 | 17
milliseconds | 255 (463) | 215 (278) | 297 (278)

2. Primary Outcome: Delay Discounting Task
Description: This task assessed discounting larger future rewards for smaller immediate ones. The point where a person is equally likely to prefer immediate vs delayed reward (the indifference point) is determined for several and combinations of reward sizes and lengths of time. Area under the curve (AUC) is calculated by summing the results of the following for each delay and indifference point pair: x2-x1[(y1 + y2)/2]. x1 and x2 are successive delays and y1 and y2 are indifference points for those delays. AUC range=0-1. Larger AUCs reflect less impulsivity.
Time Frame: Within an hour post-stimulation condition
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anodal tDCS Over the rIFG, | Anodal tDCS Over the lOFC | Sham tDCS Stimulation
Number analyzed (Participants) | 17 | 18 | 18
score on a scale | .53 (.31) | .4 (.25) | .57 (.29)

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Anodal tDCS Over the rIFG, | Anodal tDCS Over the lOFC | Sham tDCS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/20

LIMITATIONS AND CAVEATS:
Multiple and persistent technical problems were experienced with the device used in this study. It was not possible to confirm that stimulation reliably occurred and that therefore all study participants received then intended stimulation. Caution should therefore be taken in interpreting the results of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT03365102/Prot_SAP_000.pdf